CLINICAL TRIAL: NCT03065881
Title: RETeval All Comers Trial (REACT)
Acronym: REACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: LKC Technologies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: LKC-2017-1
Record Dates: First submitted 2017-02-12; First posted 2017-02-28 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Retinal Disease, Electroretinogram
MeSH Terms: conditions — Retinal Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Dilated versus Natural pupil (Active Comparator)
  Interventions: Device: RETeval
- Normal retina versus abnormal retina (Active Comparator)
  Interventions: Device: RETeval

INTERVENTIONS:
Device: RETeval — The RETeval device measures the retina's electrical response to light, called an electroretinogram (ERG). The standards body ISCEV [1] recommends collecting normative data for ERGs to provide waveforms and statistically relevant measurements representing the range of ERGs from people with normal vision. LKC Technologies provides this information with their UTAS product line and wishes to collect such a database for the newest device: the RETeval device. As the RETeval device uses a different electrode to measure the ERG, the normal data for the UTAS product line is not transferable to the RETeval device. Ophthalmic practitioners would also like ERG examples of specific retinal disorders to help diagnose patients with abnormal ERGs. The RETeval device is FDA cleared (K142567),

SUMMARY:
The primary objective of this study is to collect electroretinogram ERG measurements from visually normal and abnormal subjects using the FDA cleared RETeval device (K142567). Data from the visually normal subjects will be used to create reference intervals for the device. Secondary objectives of the study are to provide ERG waveforms representative of disease states encountered and to analyze how well an ERG detects the various disease states encountered.

ELIGIBILITY:
Inclusion Criteria:

* All volunteers (age 0.5 to 95) willing to participate in the study as a part of their routine eye exam.
* While not specifically targeting vulnerable groups such as for example children and pregnant women, we invite them to participate in the study. Collecting normative data from these less represented populations is particularly difficult and we welcome the opportunity to gather these rare data.
* Subjects under the age of 18 will be included with the assent of the subject (for those at least 10 years of age) and consent from one parent/guardian (for those under age of 10).
* In any case patient is not able to provide the consent by him/her self and is willing to participate in the study the same person that is consenting for the routine eye exam can consent for the REACT study.

Exclusion Criteria:

* Subjects with photosensitive epilepsy , allergies to pupil dilating agents, or history of cardiac dysrhythmia will not be invited to participate in this study. - Subjects with history of glaucoma can either be included in the group of non dilated subjects or can have dilated ERGs if the dilation was recommended by the health professional as the part of the routine eye exam.
* Exclusion criteria will be based on volunteer's providing this information at the time of signing the consent form.
* If patient is not aware of his photosensitive epilepsy and it occurs during the recording, the test will be interrupted immediately.
* Statistically, 1 person out of 3600 people can suffer from photosensitive epilepsy in US.
* There is a rather small possibility we will encounter such a person during the collection of ERGs from the group of 1000 volunteers

Ages: 6 Months to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 664 (Actual)
Dates: Start 2017-02-13 (Actual); Primary Completion 2021-12-21 (Actual); Study Completion 2021-12-21 (Actual)

PRIMARY OUTCOMES:
Retinal function assessed with an electroretinogram (ERG) | 1 year
  Response of the retina exposed to the flashes of light. ERG describes retinal function.

CONTACTS AND LOCATIONS:
Locations (1):
- Little Rock Eye Clinic, Little Rock, Arkansas, United States